CLINICAL TRIAL: NCT04379713
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY INFANTS
Brief Title: 20-valent Pneumococcal Conjugate Vaccine Safety Study in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B7471013; 2019-003307-35 (EudraCT Number)
Record Dates: First submitted 2020-05-06; First posted 2020-05-07 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20-valent pneumococcal conjugate vaccine (Experimental): Pneumococcal conjugate vaccine
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine
- 13-valent pneumococcal conjugate vaccine (Active Comparator): Pneumococcal conjugate vaccine
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 20-valent pneumococcal conjugate vaccine — Pneumococcal conjugate vaccine
  Arms: 20-valent pneumococcal conjugate vaccine
Biological: 13-valent pneumococcal conjugate vaccine — Pneumococcal conjugate vaccine
  Arms: 13-valent pneumococcal conjugate vaccine

SUMMARY:
This study is designed to evaluate the safety and tolerability of 20vPnC in healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants born at ≥34 weeks of gestation and who are 2 months of age (≥42 to ≤98 days) at the time of consent (the day of birth is considered day of life 1).
* Healthy infants determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study.

Exclusion Criteria:

* Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt through study participation.
* Major known congenital malformation or serious chronic disorder.

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1511 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (97):
- United States (41):
  - Eclipse Clinical Research, Tucson, Arizona
  - Good Samaritan Family Health Team, Fullerton, California
  - FocilMed, Oxnard, California
  - Superior Research, LLC, Sacramento, California
  - Carey Chronis, MD, Ventura, California
  - Fomat - Robert Nudelman MD, Westlake Village, California
  - Ebert Family Clinic, Frisco, Colorado
  - Advanced Research for Health Improvement, LLC, Fort Myers, Florida
  - Pensacola Pediatrics, Gulf Breeze, Florida
  - Y&L Advance Health Care Inc, d/b/a Elite, Miami, Florida
  - Advanced Research for Health Improvement, LLC, Naples, Florida
  - Citadelle Clinical Research, North Miami Beach, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - Pensacola Pediatrics, Pensacola, Florida
  - KIDZ Medical Services Pediatric Pulmonary Center, South Miami, Florida
  - Teena Hughes/PAS Research, Tampa, Florida
  - Idaho Falls Pediatrics, Ammon, Idaho
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - Idaho Falls Pediatrics, Idaho Falls, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - The Pediatric Center, Idaho Falls, Idaho
  - Cotton O'Neil Clinical Research Center, Pediatrics, Topeka, Kansas
  - All Children Pediatrics, Louisville, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - MedClinical Research Partners, LLC, East Orange, New Jersey
  - Advantage Clinical Trials, The Bronx, New York
  - Pediatric Partners, PA, Raleigh, North Carolina
  - PMG Research Inc., d/b/a PMG Research of Piedmont HealthCare, Statesville, North Carolina
  - Ford Simpson Lively and Rice Pedtrics, PA (Wake Health Network), Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Pediatric Research, Summerville, South Carolina
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Advent Health Family Medicine Rural Health Clinics, Inc., Lampasas, Texas
  - FMC Science, Lampasas, Texas
  - Maximos Ob/Gyn, League City, Texas
  - Rio Grande Valley Clinical Research Institute, Pharr, Texas
  - Tanner Clinic, Layton, Utah
  - Wasatch Pediatrics - St. Marks Office, Salt Lake City, Utah
  - CopperView Medical Center, South Jordan, Utah
  - PI-Coor Clinical Research LLC, Burke, Virginia
- Argentina (3):
  - Clinica Mayo UMCB S.R.L., San Miguel de Tucumán, Tucumán Province
  - Hospital del Nino Jesus, San Miguel de Tucumán, Tucumán Province
  - Centro Medico Dra. De Salvo, Buenos Aires
- Canada (8):
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Dawson Clinical Research Inc., Guelph, Ontario
  - Milestone Research , Inc, London, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Dr. Hartley Garfield Medicine Professional Corporation, Toronto, Ontario
  - Centre hospitalier universitaire (CHU) Sainte-Justine, Montreal, Quebec
  - McGill University Health Centre, Vaccine Study Centre, Pierrefonds, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
- Chile (5):
  - CESFAM Colina, Colina, Santiago, Santiago Metropolitan
  - CESFAM Esmeralda, Colina, Santiago, Santiago Metropolitan
  - Biocinetic, Santiago, Santiago Metropolitan
  - Grupo Estudios Clínicos Infectología Respiratoria, Santiago, Santiago Metropolitan
  - Hospital Padre Hurtado, Santiago, Santiago Metropolitan
- Czechia (3):
  - Ordinace praktickeho lekare pro deti a dorost, Hradec Králové
  - Ordinace praktickeho lekare pro deti a dorost, Jindrichuv Hradec II
  - Detska ambulance Petriny spol. s r.o., Veleslavín
- MeVac - Meilahti Vaccine Research Center, Helsinki, Finland
- Germany (6):
  - SIBAmed GmbH & Co.KG, Leipzig, Saxony
  - Kinderarztpraxis Bramsche, Bramsche
  - Arztpraxis Dr. med. Dr. rer. nat. Helmut Pabel, Herford
  - Praxis fuer Kinderpneumologie und Allergologie Mannheim, Mannheim
  - Kinderarztpraxis Ralph Köllges, Jacek Mossakowski, Dr. med. Martina Meyer-Krott, Mönchengladbach
  - Praxis Dr. med. Joachim Weimer, Reinfeld
- Greece (6):
  - University General Hospital of Heraklion, Heraklion, Crete
  - General University Hospital of Larissa, Larissa, Thessaly
  - "Aghia Sophia" Children's Hospital, Athens
  - P. and A. Kyriakou Children's Hospital, Athens
  - University General Hospital "ATTIKON", Athens
  - "Ippokratio" General Hospital of Thessaloniki, Thessaloniki
- Hungary (9):
  - Papp és Tsa Eü és Szolg Bt, Szigetvár, Baranya
  - Dr Pölöskey Péter Egyéni Cég Házi Gyermekorvosi Szolgálat Szombathely, Szombathely, Vas County
  - Gyerkőc Med Bt. Házi Gyermekorvosi Rendelő, Budapest
  - Futurenest Kft. Pestszentimrei Gyermekrendelő, Budapest
  - Gyorine dr Bari Eszter E. V. 1. sz. Gyermek Haziorvosi Praxis, Csongrád
  - Futurenest Kft. 16. házi gyermekorvosi rendelő, Debrecen
  - Mimiped Bt, Győr
  - Futurenest Kft, Miskolc
  - Bettimedical BT, Százhalombatta
- Ponce Medical School Foundation Inc./ CAIMED Center, Ponce, Puerto Rico
- Spain (14):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruna
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Centro de Salud de Burriana II, Burriana, Castellon
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Centro de Salud L'Eliana, L'Eliana, Valencia
  - Centro de Salud de Paiporta, Paiporta, Valencia
  - Clinica Corachan, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Grupo Pediatrico Uncibay, Málaga
  - Centro de Salud de Malvarrosa, Valencia
  - FISABIO, Valencia
  - Centro de Salud la Serreria II, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471013

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1511 participants were enrolled and randomized to receive 4 doses of 20-valent pneumococcal conjugate vaccine (20vPnC) or 13vPnC of which 7 participants were not vaccinated and 1504 were vaccinated with either 20vPnC or 13vPnC.
Groups:
- 20vPnC: Infants 42 to 98 days of age were enrolled to receive 4 doses of 0.5 milliliter (mL) 20vPnC intramuscularly. Dose 1 was given at enrollment. Dose 2 was given 42 to 63 days later. Dose 3 was given 42 to 63 days after Dose 2. Dose 4 was administered between 12 to 15 months of age.
- 13vPnC: Infants 42 to 98 days of age were enrolled to receive 4 doses of 0.5 mL 13vPnC intramuscularly. Dose 1 was given at enrollment. Dose 2 was given 42 to 63 days later. Dose 3 was given 42 to 63 days after Dose 2. Dose 4 was administered between 12 to 15 months of age.
Period: Overall Study
Arm/Group | 20vPnC | 13vPnC
Started | 1006 | 505
Dose 1 | 1000 | 504 (One participant who was randomized to 13vPnC group incorrectly received 20vPnC vaccination.)
Dose 2 | 972 | 492
Dose 3 | 964 | 483
Dose 4 | 923 | 462
Completed | 910 | 451
Not Completed | 96 | 54
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 11 | 6
Not completed — No longer met eligibility criteria | 14 | 11
Not completed — Withdrawal by parent/guardian | 36 | 15
Not completed — Lost to Follow-up | 31 | 21

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of the investigational product with safety follow up after any dose. Participant who received any incorrect study vaccination during the study was excluded.
Groups:
- 20vPnC: Infants 42 to 98 days of age were enrolled to receive 4 doses of 0.5 mL 20vPnC intramuscularly. Dose 1 was given at enrollment. Dose 2 was given 42 to 63 days later. Dose 3 was given 42 to 63 days after Dose 2. Dose 4 was administered between 12 to 15 months of age.
- Total: Total of all reporting groups
Arm/Group | 20vPnC | 13vPnC | Total
Number analyzed (Participants) | 1000 | 503 | 1503
Age, Continuous [Mean (Standard Deviation); unit: Days] | 64.6 (8.51) | 65.0 (8.95) | 64.8 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 483 | 259 | 742
  Male | 517 | 244 | 761
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 367 | 193 | 560
  Not Hispanic or Latino | 621 | 303 | 924
  Unknown or Not Reported | 12 | 7 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 21 | 10 | 31
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 55 | 15 | 70
  White | 868 | 445 | 1313
  More than one race | 35 | 21 | 56
  Unknown or Not Reported | 15 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 1
Description: Local reactions included pain at injection site, redness and swelling, recorded by parent's/legal guardians of participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device (caliper) units. 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild: greater than (>) 0.0 to 2.0 cm; moderate: >2.0 to 7.0 cm; and severe: >7.0 cm. Pain at injection site was graded as mild: hurt if gently touched; moderate: hurt if gently touched with crying; severe: limited limb movement.
Time Frame: Within 7 Days after Dose 1
Population: Safety population included all participants who received at least 1 dose of the investigational product with safety follow up after any dose. Participant who received incorrect vaccination was excluded from analysis. Here, "Number of Participants Analyzed" signifies number of participants with any e-diary data reported after Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 992 | 498
Percentage of participants
  Redness: Mild | 18.0 (15.7) [15.7 to 20.6] | 16.5 (13.3) [13.3 to 20.0]
  Redness: Moderate | 3.7 (2.6) [2.6 to 5.1] | 3.0 (1.7) [1.7 to 4.9]
  Redness: Severe | 0 (0.0) [0.0 to 0.4] | 0 (0.0) [0.0 to 0.7]
  Swelling: Mild | 13.8 (11.7) [11.7 to 16.1] | 11.2 (8.6) [8.6 to 14.4]
  Swelling: Moderate | 6.1 (4.7) [4.7 to 7.8] | 5.4 (3.6) [3.6 to 7.8]
  Swelling: Severe | 0 (0.0) [0.0 to 0.4] | 0 (0.0) [0.0 to 0.7]
  Pain at injection site: Mild | 24.8 (22.1) [22.1 to 27.6] | 25.3 (21.5) [21.5 to 29.4]
  Pain at injection site: Moderate | 15.5 (13.3) [13.3 to 17.9] | 16.7 (13.5) [13.5 to 20.2]
  Pain at injection site: Severe | 0.2 (0.0) [0.0 to 0.7] | 0 (0.0) [0.0 to 0.7]

2. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 2
Description: Local reactions included pain at injection site, redness and swelling, recorded by parent's/legal guardians of participants in an e-diary. Redness and swelling were measured and recorded in measuring device (caliper) units. 1 measuring device unit =0.5 cm. Redness and swelling were graded as mild: >0.0 to 2.0 cm; moderate: >2.0 to 7.0 cm; and severe: >7.0 cm. Pain at injection site was graded as mild: hurt if gently touched; moderate: hurt if gently touched with crying; severe: limited limb movement.
Time Frame: Within 7 Days after Dose 2
Population: Safety population included all participants who received at least 1 dose of the investigational product with safety follow up after any dose. Participant who received incorrect vaccination was excluded from analysis. Here, "Number of Participants Analyzed" signifies number of participants with any e-diary data reported after Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 952 | 485
Percentage of participants
  Redness: Mild | 20.4 (17.9) [17.9 to 23.1] | 19.4 (16.0) [16.0 to 23.2]
  Redness: Moderate | 3.2 (2.1) [2.1 to 4.5] | 3.9 (2.4) [2.4 to 6.1]
  Redness: Severe | 0 (0.0) [0.0 to 0.4] | 0 (0.0) [0.0 to 0.8]
  Swelling: Mild | 13.4 (11.3) [11.3 to 15.8] | 13.4 (10.5) [10.5 to 16.8]
  Swelling: Moderate | 4.4 (3.2) [3.2 to 5.9] | 5.6 (3.7) [3.7 to 8.0]
  Swelling: Severe | 0 (0.0) [0.0 to 0.4] | 0 (0.0) [0.0 to 0.8]
  Pain at the injection site: Mild | 20.8 (18.3) [18.3 to 23.5] | 20.2 (16.7) [16.7 to 24.1]
  Pain at the injection site: Moderate | 10.7 (8.8) [8.8 to 12.9] | 11.8 (9.0) [9.0 to 15.0]
  Pain at the injection site: Severe | 0.7 (0.3) [0.3 to 1.5] | 0.8 (0.2) [0.2 to 2.1]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 3
Description: as for outcome 2
Time Frame: Within 7 Days after Dose 3
Population: Safety population included all participants who received at least 1 dose of the investigational product with safety follow up after any dose. Participant who received incorrect vaccination was excluded from analysis. Here, "Number of Participants Analyzed" signifies number of participants with any e-diary data reported after Dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 940 | 477
Percentage of participants
  Redness: Mild | 19.4 (16.9) [16.9 to 22.0] | 17.0 (13.7) [13.7 to 20.7]
  Redness: Moderate | 3.8 (2.7) [2.7 to 5.3] | 3.1 (1.8) [1.8 to 5.1]
  Redness: Severe | 0 (0.0) [0.0 to 0.4] | 0.2 (0.0) [0.0 to 1.2]
  Swelling: Mild | 12.2 (10.2) [10.2 to 14.5] | 13.0 (10.1) [10.1 to 16.4]
  Swelling: Moderate | 4.1 (3.0) [3.0 to 5.6] | 3.1 (1.8) [1.8 to 5.1]
  Swelling: Severe | 0 (0.0) [0.0 to 0.4] | 0.2 (0.0) [0.0 to 1.2]
  Pain at the injection site: Mild | 16.3 (14.0) [14.0 to 18.8] | 16.6 (13.3) [13.3 to 20.2]
  Pain at the injection site: Moderate | 8.3 (6.6) [6.6 to 10.2] | 10.3 (7.7) [7.7 to 13.4]
  Pain at the injection site: Severe | 0.1 (0.0) [0.0 to 0.6] | 0 (0.0) [0.0 to 0.8]

4. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 4
Description: as for outcome 2
Time Frame: Within 7 Days after Dose 4
Population: Safety population included all participants who received at least 1 dose of the investigational product with safety follow up after any dose. Participant who received incorrect vaccination was excluded from analysis. Here, "Number of Participants Analyzed" signifies number of participants with any e-diary data reported after Dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 892 | 454
Percentage of participants
  Redness: Mild | 15.1 (12.8) [12.8 to 17.7] | 19.4 (15.8) [15.8 to 23.3]
  Redness: Moderate | 5.9 (4.5) [4.5 to 7.7] | 2.4 (1.2) [1.2 to 4.3]
  Redness: Severe | 0.1 (0.0) [0.0 to 0.6] | 0 (0.0) [0.0 to 0.8]
  Swelling: Mild | 10.1 (8.2) [8.2 to 12.3] | 11.5 (8.7) [8.7 to 14.7]
  Swelling: Moderate | 4.7 (3.4) [3.4 to 6.3] | 2.9 (1.5) [1.5 to 4.8]
  Swelling: Severe | 0 (0.0) [0.0 to 0.4] | 0 (0.0) [0.0 to 0.8]
  Pain at the injection site: Mild | 19.8 (17.3) [17.3 to 22.6] | 21.8 (18.1) [18.1 to 25.9]
  Pain at the injection site: Moderate | 10.2 (8.3) [8.3 to 12.4] | 10.1 (7.5) [7.5 to 13.3]
  Pain at the injection site: Severe | 0.8 (0.3) [0.3 to 1.6] | 0 (0.0) [0.0 to 0.8]

5. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 1
Description: Systemic events included fever, decreased appetite, drowsiness, and irritability. Fever was defined as temperature greater than or equal to (>=) 38.0 degrees Celsius (C) and categorized as >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0 degrees C. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability was graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted).
Time Frame: Within 7 Days after Dose 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 992 | 498
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 6.3 [4.8 to 7.9] | 7.8 [5.6 to 10.6]
  Fever: >38.4 degrees C to 38.9 degrees C | 2.3 [1.5 to 3.5] | 1.8 [0.8 to 3.4]
  Fever: >38.9 degrees C to 40.0 degrees C | 0.7 [0.3 to 1.4] | 0.2 [0.0 to 1.1]
  Fever: >40.0 degrees C | 0 [0.0 to 0.4] | 0 [0.0 to 0.7]
  Decreased appetite: Mild | 14.2 [12.1 to 16.5] | 14.7 [11.7 to 18.1]
  Decreased appetite: Moderate | 10.3 [8.5 to 12.3] | 8.6 [6.3 to 11.5]
  Decreased appetite: Severe | 0.5 [0.2 to 1.2] | 0.4 [0.0 to 1.4]
  Drowsiness: Mild | 48.5 [45.3 to 51.6] | 47.4 [42.9 to 51.9]
  Drowsiness: Moderate | 15.8 [13.6 to 18.2] | 14.5 [11.5 to 17.9]
  Drowsiness: Severe | 0.5 [0.2 to 1.2] | 0.4 [0.0 to 1.4]
  Irritability: Mild | 22.7 [20.1 to 25.4] | 22.9 [19.3 to 26.8]
  Irritability: Moderate | 41.2 [38.1 to 44.4] | 41.4 [37.0 to 45.8]
  Irritability: Severe | 4.3 [3.2 to 5.8] | 4.2 [2.6 to 6.4]

6. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2
Description: Systemic events included fever, decreased appetite, drowsiness, and irritability. Fever was defined as temperature >=38.0 degrees C and categorized as >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0 degrees C. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability was graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted).
Time Frame: Within 7 Days after Dose 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 952 | 485
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 10.6 [8.7 to 12.7] | 8.5 [6.1 to 11.3]
  Fever: >38.4 degrees C to 38.9 degrees C | 3.6 [2.5 to 5.0] | 2.7 [1.4 to 4.5]
  Fever: >38.9 degrees C to 40.0 degrees C | 1.4 [0.7 to 2.3] | 0.2 [0.0 to 1.1]
  Fever: >40.0 degrees C | 0 [0.0 to 0.4] | 0 [0.0 to 0.8]
  Decreased appetite: Mild | 13.4 [11.3 to 15.8] | 12.0 [9.2 to 15.2]
  Decreased appetite: Moderate | 9.6 [7.8 to 11.6] | 8.2 [6.0 to 11.1]
  Decreased appetite: Severe | 0.7 [0.3 to 1.5] | 0.4 [0.0 to 1.5]
  Drowsiness: Mild | 35.3 [32.3 to 38.4] | 35.3 [31.0 to 39.7]
  Drowsiness: Moderate | 13.4 [11.3 to 15.8] | 13.8 [10.9 to 17.2]
  Drowsiness: Severe | 0.4 [0.1 to 1.1] | 1.2 [0.5 to 2.7]
  Irritability: Mild | 23.2 [20.6 to 26.0] | 19.8 [16.3 to 23.6]
  Irritability: Moderate | 37.3 [34.2 to 40.4] | 42.7 [38.2 to 47.2]
  Irritability: Severe | 4.2 [3.0 to 5.7] | 5.2 [3.4 to 7.5]

7. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 3
Description: as for outcome 6
Time Frame: Within 7 Days after Dose 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 940 | 477
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 7.4 [5.9 to 9.3] | 8.2 [5.9 to 11.0]
  Fever: >38.4 degrees C to 38.9 degrees C | 2.9 [1.9 to 4.2] | 0.6 [0.1 to 1.8]
  Fever: >38.9 degrees C to 40.0 degrees C | 1.3 [0.7 to 2.2] | 1.0 [0.3 to 2.4]
  Fever: >40.0 degrees C | 0 [0.0 to 0.4] | 0 [0.0 to 0.8]
  Decreased appetite: Mild | 15.0 [12.8 to 17.4] | 10.5 [7.9 to 13.6]
  Decreased appetite: Moderate | 8.2 [6.5 to 10.1] | 6.3 [4.3 to 8.9]
  Decreased appetite: Severe | 0.4 [0.1 to 1.1] | 0.4 [0.1 to 1.5]
  Drowsiness: Mild | 26.6 [23.8 to 29.5] | 27.3 [23.3 to 31.5]
  Drowsiness: Moderate | 8.5 [6.8 to 10.5] | 9.0 [6.6 to 12.0]
  Drowsiness: Severe | 0.2 [0.0 to 0.8] | 0 [0.0 to 0.8]
  Irritability: Mild | 22.3 [19.7 to 25.1] | 22.2 [18.6 to 26.2]
  Irritability: Moderate | 30.1 [27.2 to 33.2] | 29.8 [25.7 to 34.1]
  Irritability: Severe | 2.3 [1.5 to 3.5] | 2.7 [1.5 to 4.6]

8. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 4
Description: as for outcome 6
Time Frame: Within 7 Days after Dose 4
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 892 | 454
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 9.8 [7.9 to 11.9] | 9.5 [6.9 to 12.5]
  Fever: >38.4 degrees C to 38.9 degrees C | 4.5 [3.2 to 6.1] | 4.2 [2.5 to 6.5]
  Fever: >38.9 degrees C to 40.0 degrees C | 3.7 [2.6 to 5.2] | 3.1 [1.7 to 5.1]
  Fever: >40.0 degrees C | 0.1 [0.0 to 0.6] | 0.2 [0.0 to 1.2]
  Decreased appetite: Mild | 16.1 [13.8 to 18.7] | 12.3 [9.5 to 15.7]
  Decreased appetite: Moderate | 10.5 [8.6 to 12.7] | 11.7 [8.9 to 15.0]
  Decreased appetite: Severe | 1.7 [0.9 to 2.8] | 1.8 [0.8 to 3.4]
  Drowsiness: Mild | 24.2 [21.4 to 27.2] | 25.1 [21.2 to 29.4]
  Drowsiness: Moderate | 12.2 [10.1 to 14.6] | 10.6 [7.9 to 13.8]
  Drowsiness: Severe | 0.7 [0.2 to 1.5] | 0.2 [0.0 to 1.2]
  Irritability: Mild | 21.4 [18.8 to 24.3] | 22.0 [18.3 to 26.1]
  Irritability: Moderate | 31.4 [28.4 to 34.5] | 29.7 [25.6 to 34.2]
  Irritability: Severe | 2.5 [1.6 to 3.7] | 3.3 [1.9 to 5.4]

9. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Dose 1 to 1 Month After Dose 3
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From Dose 1 to 1 Month after Dose 3
Population: Safety population included all participants who received at least 1 dose of the investigational product with safety follow up after any dose. Participant who received incorrect vaccination was excluded from analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 1000 | 503
Percentage of participants | 29.6 (26.8) [26.8 to 32.5] | 27.6 (23.8) [23.8 to 31.8]

10. Primary Outcome: Percentage of Participants With AEs From Dose 4 to 1 Month After Dose 4
Description: as for outcome 9
Time Frame: From Dose 4 to 1 Month after Dose 4
Population: Safety population included all participants who received at least 1 dose of the investigational product with safety follow up after any dose. Participant who received incorrect vaccination was excluded from analysis. Here, "Number of Participants Analyzed" signifies number of participants who received Dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 923 | 461
Percentage of participants | 15.1 (12.8) [12.8 to 17.5] | 15.8 (12.6) [12.6 to 19.5]

11. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Dose 1 to 6 Months After Dose 4
Description: A SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/incapacity; congenital anomaly/birth defect and other important medical events.
Time Frame: From Dose 1 to 6 Months after Dose 4
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 1000 | 503
Percentage of participants | 4.4 (3.2) [3.2 to 5.9] | 5.6 (3.7) [3.7 to 7.9]

12. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) From Dose 1 to 6 Months After Dose 4
Description: An NDCMC was defined as a significant disease or medical condition, not previously identified, that is expected to be persistent or was otherwise long-lasting in its effects.
Time Frame: From Dose 1 to 6 Months after Dose 4
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 1000 | 503
Percentage of participants | 2.8 (1.9) [1.9 to 4.0] | 2.8 (1.5) [1.5 to 4.6]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events recorded using systematic assessment: within 7 days after Dose 1, 2, 3, 4; SAEs and all-cause mortality recorded using non-systematic assessment: From Dose 1 up to 6 months after Dose 4; other AEs recorded using non-systematic assessment: from Dose 1 up to 1 month after Dose 3 and from Dose 4 up to 1 month after Dose 4
Description: The same event may appear as both AE and SAE. However, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Safety population included all participants who received at least 1 dose of the investigational product with safety follow up after any dose. Participant who received incorrect vaccination was excluded from analysis.
Arm/Group | 20vPnC | 13vPnC
All-Cause Mortality (participants affected / at risk) | 0/1000 | 0/503
Serious Adverse Events (participants affected / at risk) | 44/1000 | 28/503
Other Adverse Events (participants affected / at risk) | 960/1000 | 481/503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20vPnC (N=1000) | 13vPnC (N=503)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Allergic colitis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Adverse food reaction (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 3
Anaphylactic reaction (Immune system disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Adenovirus infection (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 5 | 5
Bronchitis (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 1 | 1
Croup infectious (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 2
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 2
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Viraemia (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
Infantile spasms (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Breath holding (Psychiatric disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 20vPnC (N=1000) | 13vPnC (N=503)
Injection site erythema (REDNESS) (General disorders) | 455 | 224
Injection site pain (PAIN) (General disorders) | 609 | 309
Injection site swelling (SWELLING) (General disorders) | 372 | 176
Pyrexia (FEVER) (General disorders) | 336 | 159
Upper respiratory tract infection (Infections and infestations) | 59 | 28
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 549 | 249
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 809 | 389
Irritability (IRRITABILITY) (Psychiatric disorders) | 883 | 432

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT04379713/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT04379713/SAP_001.pdf